CLINICAL TRIAL: NCT06246058
Title: Measuring Anticipated Attitudes and Behavior Towards a New Medical Treatment in Lesotho
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: SolidarMed (Other)
Responsible Party: Sponsor
Other Study IDs: ID213-2023; ub23Belus
Record Dates: First submitted 2024-01-08; First posted 2024-02-07 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Health Behavior; Motivation; Health Care Utilization; Consumer Behavior; Social Behavior; Health Care Seeking Behavior; Recruitment; Researcher-Subject Relations
Keywords: Social support; Uncertainty; Low-resource setting; Ambiguity aversion; Behavioral economics; Research administration; Recruitment success
MeSH Terms: conditions — Health Behavior; Patient Acceptance of Health Care; Consumer Behavior; Social Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Survey Group 1 - Support: Receives a vignette with partner support component before answering AA-Med response items.
  Interventions: Behavioral: Partner support
- Survey Group 2 - Control: Receives a vignette without partner support component before answering AA-Med response items.
  Interventions: Behavioral: Without Partner support
- Recruitment Group 1 - Casual: Recruited by staff wearing casual attire.
  Interventions: Behavioral: Casual recruiter attire
- Recruitment Group 2 - Formal: Recruited by staff wearing formal (clinical) attire
  Interventions: Behavioral: Formal recruiter attire

INTERVENTIONS:
Behavioral: Partner support — The intervention group's survey vignette will include a component of partner support which serves as the key behavioral manipulation tested for this study's primary outcome.
  Groups: Survey Group 1 - Support
Behavioral: Formal recruiter attire — The SWAT will separately test recruitment rates - as measured by rate of survey completion divided by total number of individuals approached - based on how the recruiters are dressed.
  FORMAL dress code of the recruiter is the intervention in this case, defined as clinical attire alluding to some clinical authority.
  Groups: Recruitment Group 2 - Formal
Behavioral: Without Partner support — The intervention group's survey vignette will NOT include a component of partner support which serves as the key behavioral manipulation tested for this study's primary outcome.
  Groups: Survey Group 2 - Control
Behavioral: Casual recruiter attire — The SWAT will separately test recruitment rates - as measured by rate of survey completion divided by total number of individuals approached - based on how the recruiters are dressed.
  CASUAL dress code of the recruiter is the intervention in this case.
  Groups: Recruitment Group 1 - Casual

SUMMARY:
The primary research objective is to examine how uncertainty towards a new medical treatment changes in patients when a partner (can be any close other, i.e. romantic partner, family member, or a close friend) supports the new treatment choice and is willing to be involved in the patient's treatment. I hypothesize that when the patients know that their partner supports uptake of the new medical treatment and will physically accompany them to the visit, patients will (1) experience lower levels of uncertainty and (2) report a higher likelihood of participating in a new treatment in the future, as compared to patients who face the decision about the new treatment alone.

DETAILED DESCRIPTION:
Host trial: Uncertainty survey experiment

This study uses a survey experiment with a hypothetical scenario (vignette) to test the concept of uncertainty and the impact of partner involvement in a hypothetical new medical treatment in patients seeking healthcare in the Butha Buthe district hospital. Specifically, this host trial will be a single-blinded randomized survey experimental design. This means that there will be two versions of the vignette and participants will be randomly given only one version (1:1 allocation). The participants will not be made aware that there is a different version of the vignette but the researchers will be aware of which version the participant receives. The difference between the vignettes (called behavioral manipulation) is whether or not the partner endorses the hypothetical new medical treatment related to the patient's current illness. See the Study measures Section for the specific vignettes.

Study Within a Trial (SWAT): Impact of the researcher's attire on recruitment rates

Within the host trial, the nested study on researcher's attire will take place as a "Study Within A Trial" or SWAT. SWAT is an increasingly recognized method of research that aims to improve the research methodology within an existing trial. The SWAT on researcher attire will take place in the recruitment phase of the host experiment with day-based cluster randomization between white coat versus casual attire assignment. These attire assignments will be given along with the given week's recruitment assignments to the two Basotho research assistants who will work on the host trial. The nested study does not impact the procedures of the survey experiment. Researcher's attire during recruitment will remain the same throughout the survey delivery until the end of the participant's study visit.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age
* Are comfortable reading and writing in Sesotho or English
* Attending as a patient in Butha Buthe-area hospital or health center for a known clinical diagnosis or standard health screening related to one of these illness categories:
* HIV
* Other sexually-transmitted infection (i.e. gonorrhea, syphilis, hepatitis)
* Breathing problem/ tuberculosis
* Heart issues/ blood pressure
* Diabetes/ sugar level
* Bone/ muscle problem
* Mental health
* Memory/ thinking problem
* Teeth/ mouth problem
* Cancer
* Maternal health (i.e. pregnancy, post-partum care)

Exclusion Criteria:

* Have participated in this study before
* Visible intoxication and/or distress, as deemed by trained research assistant
* Unable to make independent decisions; unable to complete informed consent
* Warrants emergency medical care
* Visiting the hospital for another person (i.e. their child, relative, partner)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruitment will occur in the Butha Buthe district hospital and health centers in the Butha Buthe district.
Sampling Method: Probability Sample
Enrollment: 475 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-09-13 (Actual)

PRIMARY OUTCOMES:
AA-Med score | 1 time measurement immediately after intervention
  Ambiguity aversion score difference between two survey groups; AA-Med contains 6 response items, each scored from 1 to 4 (1=disagree completely; 4=agree completely)

SECONDARY OUTCOMES:
Recruitment rate | 1 time measurement immediately after intervention
  Recruitment success rate (fully participated/ approached) difference between two recruitment attire groups

CONTACTS AND LOCATIONS:
Overall Officials: Grace H Yoon, MSc, Principal Investigator — University Hospital Basel, University of Basel
Locations (1):
- Butha Buthe Government Hospital, Butha-Buthe, Lesotho

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest. Data shared will be completely anonymized. Study components, aggregate data and results will be disseminated on OSF. Any additional data sharing is subject to approval of the request and execution of all applicable agreements (i.e. a material transfer agreement).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting six months after completion of data collection for up to 24 months thereafter.
Access Criteria: Independent researchers with academic interest.
URL: https://osf.io/mvkqc/?view_only=643a466e48d6433586d275e2f15f2770

REFERENCES:
- [Background] Han PK, Reeve BB, Moser RP, Klein WM. Aversion to ambiguity regarding medical tests and treatments: measurement, prevalence, and relationship to sociodemographic factors. J Health Commun. 2009 Sep;14(6):556-72. doi: 10.1080/10810730903089630. PMID 19731127
- See also: OSF project page — https://osf.io/mvkqc/?view_only=643a466e48d6433586d275e2f15f2770